CLINICAL TRIAL: NCT03736941
Title: Impact of Venotrain UlcerteC Venous Compression Device in the Treatment of Venous Ulcers in Daily Practice
Acronym: INVICTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INVICTUS
Record Dates: First submitted 2018-11-05; First posted 2018-11-09 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with venous leg (Experimental): After inclusion, the medical device Venotrain® Ulcertec will be prescribed according to the indications supported by the Health Insurance and used according to the recommendations of the manufacturer. Follow-up visits are scheduled at 4, and 16 weeks (± 1 week) as well as an end-of-study visit, not later than 20 weeks after enrollment or in case of premature termination. follow-up.
  During the various visits, clinical data will be collected in the patient's medical file as well as the answers to the questionnaires.
  Interventions: Other: Patients with venous leg

INTERVENTIONS:
Other: Patients with venous leg — The medical device Venotrain® Ulcertec will be prescribed according to the indications supported by the Health Insurance and used according to the recommendations of the manufacturer. It will be dispensed in town pharmacies. After inclusion, follow-up visits are scheduled at 4, and 16 weeks (± 1 week) as well as an end-of-study visit, not later than 20 weeks after enrollment or in case of premature termination. follow-up.

SUMMARY:
The cornerstone of the management of venous leg or predominantly venous leg ulcers with IPS> 0.8 is venous compression as recommended by the HAS in June 2006. There is ample clinical evidence to support its importance to improve the chances of closure of this chronic lesion and shorten the healing time compared to the absence of compression.

In 2016, a system of re-usable compression stockings (Venotrain® Ulcertec, BAUERFEIND, France), and bringing an interface pressure of 30 to 45 mmHg to the ankle according to the prescription, was taken over by the Health Insurance in France. 'Indication' Ulcer of venous origin or predominantly venous component, stage C6 CEAP classification with a systolic pressure index greater than 0.9 '.

The investigators propose to study the efficiency of Venotrain® Ulcertec in a diverse population in which it is prescribed according to the usual practices of venous leg ulceration of venous or predominantly venous origin.

DETAILED DESCRIPTION:
The supra-malleolar leg ulcers of venous origin, in the C6 stage of the CEAP (unhealed venous ulcer), are characterized by the presence of two pulses (pedis and posterior tibial) or a Systolic Pressure Index (SPI) ≥ 0, 7 or a pressure of the big toe ≥ 60 mmHg or an arterial echo-doppler of the lower limbs revealing neither hemodynamic stenosis nor arterial occlusion.

The HAS working group defines a pure venous ulcer as a leg wound that has not healed for more than 1 month, related to an ambulatory venous hyperpressure. This hyperpressure may be secondary to superficial vein reflux and / or deep vein reflux or obstruction and / or calf pump deficiency. In the pure venous ulcer, there is no arterial involvement. The predominantly venous mixed ulcer is an ulcer with a preferentially venous mechanism but accompanied by a moderate arterial occlusion of the lower limbs which does not explain the symptomatology alone.

The fundamental element in the management of venous or predominantly venous leg ulcers with an SPI> 0.8 is venous compression as recommended by the June 2006 HAS.

Numerous clinical evidence confirms its importance for improving the chances of closure of this chronic lesion and shortening the healing time compared to the absence of compression.

It is a long treatment that can last several months, very restrictive for the patient and all the more so, that the perception of an improvement is far from immediate. In addition, the affected population is usually elderly, and the ulcer is a source of permanent discomfort, affecting the quality of life of the subjects and explaining frequent social isolation and depressed mood. Moreover, the cost of this treatment is sometimes dissuasive with a dependent burden for the patient who, sometimes, is unacceptable.

In 2016, a system of re-usable compression stockings (Venotrain® Ulcertec, BAUERFEIND, France), and bringing an interface pressure of 30 to 45 mmHg to the ankle according to the prescription, was taken over by the Health Insurance in France. 'indication' Ulcer of venous origin or predominantly venous component, stage C6 of the CEAP classification (ie not healed) with a systolic pressure index greater than 0,9 '. This type of device has demonstrated an efficiency of the same order as the multi-type or multi-band systems for the closure of venous ulcers.

The investigators can therefore hope for the use of this type of stockings, a simplification of the care, an improvement of the comfort of wearing and thus a reduction of the feeling of frustration on the part of the patients with main consequence a better acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with venous or predominantly venous leg ulcer as defined by HAS
* Patient with at least one supracleolar ulcer at stage C6 of CEAP
* Surface of the ulcer of the largest size ≤ 10 cm2
* IPS less than 6 months> 0.8 for both limbs or toe pressure ≥ 60 mmHg if mediacalcosis (SPI> 1.2)
* Patient with a maximum of three supraballeolar ulcers (one or two sided)
* Patient followed by a hospital outpatient clinic in the departments of vascular medicine, angiology, internal medicine, dermatology or geriatric medicine (First consultation or not)
* Patient with walking ability over 50 m (with or without help)
* Patient with a prescription indication of Venetrain® Ulcertec Low Venous Compression System (Bauerfeind)
* Patient giving free, informed and written consent

Exclusion Criteria:

* Any other non-venous etiology of the ulcer in the opinion of the clinician
* Infections of lesions requiring the introduction of systemic antibiotic therapy
* Contraindication to treatment including venous compression by stockings
* Patient with cognitive impairment
* Patient to be hospitalized within 20 weeks after inclusion
* Patient with another wound than the leg ulcer (s) (especially foot ulcers, pressure ulcers)
* Patient with at least one very exudative ulcer, requiring the placement of a thick absorbent primary dressing incompatible with the use of compression stockings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Optimal efficiency | Week 20
  The primary endpoint is the overall, center-level prevalence of optimal VENOTRAIN® Ulcertec compressive sock efficiency. Optimal efficiency is defined by the observation of an ulcer closure at the end of a maximum follow-up of 20 weeks without the need to change the type of compression system initially prescribed and without detecting local problems considered by the clinician as possibly related to the compressive device but not interfering with the patient's management.

SECONDARY OUTCOMES:
health-related quality of life EQ5D-5L | Week 4
  The patient will complete the questionnary during the 4 weeks's consultation. EQ-5D is a standardized instrument for measuring generic health status.The number of levels of severity was increased to five in this new version; having no problems, having slight problems, having moderate problems, having severe problems and being unable to do/having extreme problems.
health-related quality of life EQ5D-5L | Week 16
  The patient will complete the questionnary during the 16 weeks's consultation. EQ-5D is a standardized instrument for measuring generic health status.The number of levels of severity was increased to five in this new version; having no problems, having slight problems, having moderate problems, having severe problems and being unable to do/having extreme problems.
health-related quality of life EQ5D-5L | Week 20
  The patient will complete the questionnary during the 20 weeks's consultation. EQ-5D is a standardized instrument for measuring generic health status.The number of levels of severity was increased to five in this new version; having no problems, having slight problems, having moderate problems, having severe problems and being unable to do/having extreme problems.
Prevalence of acceptable efficiency | Week 20
  The endpoint is the overall, center-level prevalence of acceptable VENOTRAIN® Ulcertec compressive sock efficiency. An acceptable efficiency will be defined according to the same criteria but at least one troublesome local event has been detected without requiring a temporary or permanent interruption of the compression system initially prescribed.
Evaluation of the patient's adhesion of VENOTRAIN® Ulcertec compressive sock | Week 4
  If stop: frequency of use before stop (never, episodic, daily), date of stop, person having decided the stop, reason for stop, prescription of another system If current use: time of use, membership (daily wear, every other day or more, less than every other day, from time to time or never / almost), ease of use of the compression according to the Likert scale, overall acceptability of Likert scale compression
Evaluation of the patient's adhesion of VENOTRAIN® Ulcertec compressive sock | Week 16
  If stop: frequency of use before stop (never, episodic, daily), date of stop, person having decided the stop, reason for stop, prescription of another system If current use: time of use, membership (daily wear, every other day or more, less than every other day, from time to time or never / almost), ease of use of the compression according to the Likert scale, overall acceptability of Likert scale compression
Evaluation of the patient's adhesion of VENOTRAIN® Ulcertec compressive sock | Week 20
  If stop: frequency of use before stop (never, episodic, daily), date of stop, person having decided the stop, reason for stop, prescription of another system If current use: time of use, membership (daily wear, every other day or more, less than every other day, from time to time or never / almost), ease of use of the compression according to the Likert scale, overall acceptability of Likert scale compression
Time's estimation to obtain complete closure | Week 20
  Time's estimation to obtain complete closure : Kaplan Meier Method

CONTACTS AND LOCATIONS:
Overall Officials: Audrey P STANSAL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Centre hospitalier universitaire d'Angers, Angers
  - Groupe Hospitalier Paris Saint-Joseph, Paris

IPD SHARING:
Plan to Share IPD: Undecided